CLINICAL TRIAL: NCT06295289
Title: Hybrid Closed-loop Insulin Delivery System in Perioperative Diabetic Patients: an Open-label, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Professor, Chief Physician，Director of Department of Endocrinology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZRKY-2023-04
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid closed-loop insulin delivery system group (Experimental): After patients signed the informed consent form in the ward, the nurse installed the insulin pump and the subcutaneous, real-time, continuous glucose monitor (CGM). The insulin pump was installed in the abdomen or upper arm, and the CGM was installed in the upper arm. A Hybrid closed-loop insulin delivery system with an open-source algorithm was set up for participants by the clinical trial investigators. The algorithm was initialized with the participant's weight and basal insulin requirements. The control algorithm modulated insulin delivery every 5 min based on the CGM glucose level, anticipated glucose trends, and patient-specific information such as the basal rate profile to guarantee blood glucose control within the target range. The perioperative patients in the hybrid closed-loop insulin delivery group who were admitted to the hospital received 3-5 days of glucose-lowering therapy.
  Interventions: Device: Hybrid Closed-loop Insulin Delivery System
- Insulin pump therapy group (Control group) (Placebo Comparator): The insulin treatment with a pump and CGM was applied according to the local clinical guidelines. The insulin pump was installed in the abdomen or upper arm, and the CGM was inserted in the upper arm by the investigator. Doctors adjust the insulin dose according to the patient's glucose level.
  Interventions: Device: Insulin pump

INTERVENTIONS:
Device: Hybrid Closed-loop Insulin Delivery System — The Hybrid Closed-loop Insulin Delivery System system consisted of a Medtronic pump, a continuous glucose monitoring system（SIBIONICS®）and an open-source algorithm integrated into the phone. Insulin pump therapy group consisted of a Medtronic pump, and a continuous glucose monitoring system（SIBIONICS®). The difference between the two groups is that the artificial pancreas system automatically regulates the basal rate to maintain blood glucose in a target range.
  Arms: Hybrid closed-loop insulin delivery system group
Device: Insulin pump — Participants used conventional insulin pumps to control blood glucose, At the same time, a continuous glucose monitoring system was used to monitor glucose changes. Health care providers adjust the insulin dose of patients according to their blood glucose level.
  Arms: Insulin pump therapy group (Control group)

SUMMARY:
Perioperative management of glucose levels remains challenging. The purpose of the study is to compare the hybrid closed-loop insulin delivery system with the standard insulin therapy ( insulin pump with CGM, insulin dose controlled by physicians) in controlling glucose levels among patients in the perioperative period.

DETAILED DESCRIPTION:
Hyperglycemia is particularly frequent in the perioperative period, which leads to metabolic and functional disorders, aggravates organ damage, induces various complications, and increases the risk of postoperative infection and even death.

However, glucose level management among perioperative patients remains challenging because of the frequent blood glucose monitoring requirement and insulin adjustment to accommodate the physiological changes of patients before surgery.

In this study, we planned to use an open-source, hybrid closed-loop insulin delivery system and common insulin pump combined with CGM for short-term intensive insulin therapy in patients with diabetes during the perioperative period. To comprehensively evaluate the clinical efficacy and safety of the hybrid closed-loop insulin delivery system, we planned to compare the blood glucose control and other clinical indicators such as postoperative complications of patients with different intensive insulin therapy regimens If the participant is enrolled before the surgery, the following procedure will be followed:

Preoperative: the participants wear the open-source AP system for treatment.

Intraoperative: participants should discontinue the insulin pump in advance, with the specific timing determined by the endocrinologist. The CGM can remain in place as long as it does not interfere with the surgery.

Postoperative: After the subject returns to the ward, the nurse will reinstall the open-source AP system, and the treatment will continue for at least 3-4 days.

ELIGIBILITY:
Inclusion Criteria:

1）18~75 years old (including 18 years old and 75 years old),

2）Perioperative patients with need diabetes including type 2 diabetes mellitus and other special types of diabetes mellitus and need insulin therapy;

3）Fasting blood glucose ≥7.0mmol/L or random blood glucose 11.1≥mmol/L;

4）Patients signed the informed consent form and volunteered to participate in the clinical trial.

5 ) Patients who have already undergone surgery and are still hospitalized during the perioperative period with poor glycemic control.

Exclusion Criteria:

1. The patients were complicated with diabetic emergencies, such as diabetic ketoacidosis, diabetic hyperosmolar non-ketotic coma, etc.
2. Type 1 diabetes mellitus
3. Patients with severe cardiac and renal organ dysfunction: cardiac function above grade III; Serum creatinine over 442μmol/L; Hemoglobin less than 90g/L; White blood cell count <4.0×109/L or platelet count <90×109/L;
4. Patients who are allergic to drugs specified in clinical protocols
5. Patients who are not suitable for conventional insulin pump therapy.
6. Patients who are allergic constitution and allergic to tape
7. Patients with skin diseases such as rash and prurigo, or abnormal coagulation function;
8. Patients who suffer from mental illness, have no self-control, and cannot express themselves clearly.
9. Other circumstances that investigator considered to be inappropriate for clinical trial participation;

10) Patients with severe complications during or after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
TIR | 5-10days
  time in range

SECONDARY OUTCOMES:
TAR | 5-10days
  time above range
TBR | 5-10days
  time blow range
MBG | 5-10days
  mean blood glucose

OTHER OUTCOMES:
postoperative infection | 5-10days
  rate of postoperative infection in the perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No